CLINICAL TRIAL: NCT01686685
Title: Study of Correlation Between Expression of Proteins That Are Essential for Embryonic Brain Development and Neurodevelopmental Outcomes at 2 Years of Age in Premature Infants.
Brief Title: Correlation of CXCR4 Expression in Premature Infants With a Diagnosis of Autism at 24 Months
Acronym: ASD-CXCR4
Status: Completed | Type: Observational
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Sponsor
Other Study IDs: begin1HMO-CTIL
Record Dates: First submitted 2012-09-13; First posted 2012-09-18 (Estimated); Last update posted 2018-04-12 (Actual); Status verified 2012-09

CONDITIONS: Autism Spectrum Disorder; Complication of Prematurity
Keywords: ASD; autism; prematurity; oxygen-dependant gene activation; CXCR4; Language delay; Cognitive delay
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder; Premature Birth; Language Development Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood samples. expression of proteins or RNA will be determined from the blood.
Oversight: Data Monitoring Committee: No

SUMMARY:
Preterm children are at increased risk for autism spectrum disorders, with an estimated rate of 10%. In the US, about 1 in 8 pregnancies ends with a premature birth. Therefore, individuals with ASD who were born prematurely form a substantial body of children diagnosed with ASD.

Premature birth confers an insult to the newborn at a neurologically vulnerable stage. Prematurity associated changes in oxygen tension can be detrimental to developing organs, the brain being one of the most rapidly developing organs in the second half of the pregnancy. Changes in oxygen tension mediate activation of proteins that change the course of cell development.

In this study, we plan to measure changes in the expression of 3 proteins that may be affected by changes in oxygen level at birth. We will study the interaction between the proteins' levels in the first few days after premature birth with a diagnosis of ASD at 2 years of age. The proteins are:

1. VEGF (Vascular Endothelial Growth Factor), a protein that takes part in creating new blood vessels during embryonic development.
2. Hypoxia-inducible factor -1(HIF-1), a key protein that coordinates expression of different genes, many with developmentally critical functions.
3. CXCR4, a cell surface protein that is activated by SDF-1. SDF- 1 is a molecule that regulates migration of cells to their target destination during embryonic life. CXCR4 is expressed in areas of the brain and on cells that are known to be associated with ASD.

We hypothesis that changes in oxygen tension in premature babies initiates a cascade of events that lead to changes in cell mobility via abnormal CXCR4 expression. This change leads to abnormal neurodevelopment.

The investigators' primary aim is to find if there is a correlation between postnatal levels of expression of HIF-1, CXCR4 and VEGF and a diagnosis of autism at age 24 months. The investigators' secondary aim is to find if there is a correlation between postnatal levels of expression of HIF-1, CXCR4 and VEGF and a language or neurocognitive delay.

Methods:

1. Premature babies will be recruited in the first day post delivery.
2. Blood samples will be collected at 3 time points during their hospitalization, and the expression of HIF-1, CXCR4 and VEGF will be determined.
3. Infants will undergo a complete developmental evaluation at 18-24 months of age .
4. Postnatal levels of HIF, CXCR4 and VEGF will be plotted against the results of the developmental evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Parents gave informed consent approved by the Institutional Review Board
* Gestational week 28-34 as determined by an ultrasound during the first trimester
* Singleton or twin pregnancy

Exclusion Criteria:

* Major anatomical abnormalities as detected on prenatal US
* Genetic syndrome as detected by prenatal US, MRI or chorioamniocentesis
* Obvious anatomical abnormalities or dysmorphic features detected on physical examination immediately following birth
* Triplet pregnancy
* Mother known or suspected to consume alcohol or illegal drugs during pregnancy
* Mother took medications during pregnancy that are known to have adverse affects on development (e.g. anti-epileptics)
* Family history of genetic syndrome related to developmental delays, that was not ruled out during current pregnancy (e.g. sibling with Tuberous Sclerosis or fragile X)

Ages: 1 Hour to 1 Day | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: neonatal intensive care units newborn ward
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2013-09; Primary Completion 2018-04 (Actual); Study Completion 2018-04-01 (Actual)

PRIMARY OUTCOMES:
Diagnosis of ASD at 24 months corrected age | 30 months
  Participants will be screened at 18 and 24 months for autism using the MCHAT questionnaire all positive screens will be referred for a complete developmental evaluation by child psychologist and developmental pediatrician: History, assessment (ADOS) and clinical judgement based on DSM criteria

SECONDARY OUTCOMES:
Language or cognitive delay at 24 months corrected age | 30 months
  Participants will be screened by questionnaires at 18 and 24 months. all positive screens will be referred for a full developmental evaluation using the Mullen Scales of Early learning

CONTACTS AND LOCATIONS:
Overall Officials: Michal Begin, MD, Study Director — Hadassah HMO
Locations (1):
- Hadassah Medical Center, Jerusalem, Israel